CLINICAL TRIAL: NCT02697994
Title: Intradermal Sterile Water Injections for Labour Pain: A Randomised Controlled Trial
Brief Title: Sterile Water Injections For Pain Relief İn Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, refika genç koyucu, assist.prof., University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SWI1315
Record Dates: First submitted 2016-02-09; First posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Labour Pain; Back Pain
Keywords: Sterile Water Injection; Midwifery
MeSH Terms: conditions — Labor Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sterile Water Injection (Experimental): Participants randomised to the intervention group received 4 intracutaneous injections of 0.1 ml sterile water into the skin surrounding the Michaelis rhomboid over the sacral area.
  Interventions: Other: Sterile Water
- Dry Injection (Placebo Comparator): Participants in the control group received 4 dry injections in the same region using an insulin needle .
  Interventions: Other: Dry Injections

INTERVENTIONS:
Other: Sterile Water — 0.1 ml intracutaneous sterile water injections into the skin surrounding the Michaelis rhomboid over the sacral area.
  Arms: Sterile Water Injection
Other: Dry Injections — dry injections into the skin surrounding the Michaelis rhomboid over the sacral area.
  Arms: Dry Injection

SUMMARY:
ABSTRACT Introduction: In addition to pain caused by uterine contractions in labour, in 33% of women, continuous and severe back pain is observed. In management of this pain, sterile water injection is considered to be an effective method. Aim of this study is assessment of effectiveness and satisfaction of this method among Turkish women in which analgesic methods are not extensively used in labour and rates of cesarean section exponentially increases.

Material and Methods: 168 termed, healthy women who admitted to Istanbul Gaziosmanpaşa-Taksim Training and Research Hospital with labour pain and had severe back pain were randomized into 4x0.1 ml sterile water and 4xdry Injection groups. Injections were applied to Michaelis Rhomboid region in sacral region. Pain scores were assessed at 10th, 30th, 60th, 120th and 180th minutes with Visual Analog Scale (VAS). Additionally, need for epidural analgesia, APGAR score, mode of delivery, time of delivery, maternal satisfaction and breastfeeding scores were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35
* 37-42 weeks of gestation
* Expecting vaginal delivery
* Cephalic presentation
* Single, healthy fetus
* Spontaneous onset of labor
* Active phase of first stage of labor (3-7 cm cervical dilatation)
* Severe low back pain (VAS>7cm)
* Required pain relief

Exclusion Criteria:

* Gestation <37 weeks
* Multiple pregnancy
* Malpresentation
* Second stage labour
* Pharmacological analgesia prior to SWI
* Back pain assessed by VAS <7
* Women whose labour would be considered high risk

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pain scores-30 | at 30 mins after interventions
  In pain scoring Visual Analog Scale was used

SECONDARY OUTCOMES:
Pain scores-10 | at 10 mins after interventions
  In pain scoring Visual Analog Scale was used
Pain scores-60 | at 60 mins after interventions
  In pain scoring Visual Analog Scale was used
Pain scores-90 | at 90 mins after interventions
  In pain scoring Visual Analog Scale was used
Pain scores-120 | at 120 mins after interventions
  In pain scoring Visual Analog Scale was used
Pain scores-180 | at 180 mins after interventions
  In pain scoring Visual Analog Scale was used
APGAR score of neonate | at 5 mins after birth
Maternal satisfaction | at 1 hour after birth
  Likelihood to use again with subsequent labour, Women satisfaction with analgesic effect, Likelihood to recommend to SWI to others
Rates of breastfeeding-1 | at 1 hour after birth
  In breastfeed scoring The Infant Breastfeeding Assessment Tool was used
Rates of breastfeeding-24 | at 24.hours after birth
  In breastfeed scoring The Infant Breastfeeding Assessment Tool was used

IPD SHARING:
Plan to Share IPD: Undecided